CLINICAL TRIAL: NCT01538654
Title: Enteroprotein Modified Fast ( EMF ) : Clinical Safety and Efficacy. A Six Months Pilot RCT
Brief Title: Enteroprotein Modified Fast ( EMF )
Acronym: EMF
Status: Completed | Type: Observational
Sponsor: M.D. Samir G. Sukkar (Other)
Collaborators: Nestlé Foundation (Other)
Responsible Party: Sponsor-Investigator, M.D. Samir G. Sukkar, Chief Clinical Nutrition Unit, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Organization: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Other Study IDs: EMF2011
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: obesity; PSMF ( protein sparing modified fast); Enteral nutrition; Tube feeding; VLCD ( very low calorie diet); Pulmonary function tests; body composition; FFM ( fat free mass); Body fat; Handgripstregth
MeSH Terms: conditions — Obesity | interventions — Adiposity; Electromagnetic Fields

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 'enteral protein tube feeding in obese: protein sparing modified fast with a defined enteral formula by tube
  Interventions: Procedure: enteral protein tube feeding in obese

INTERVENTIONS:
Procedure: enteral protein tube feeding in obese — The intervention is represented by a new alternative to treat obese patients by means of a protein sparing modified fast administered by continous 24 h enteral feeding
  Other Names: EMF ( enteral modified fast )

SUMMARY:
The purposes of the esperience is:

1. to verify the safety of protein sparing modified fast(PSMF) by enteral route ( EMF )performed in cycles of ten days/months for six months
2. to compare EMF with oral PSMF clinically ( appetite control, fat freemass mantainance, polmonary function tests and metabolic pattern)
3. to verify the weight mantainance after 6 months from the treatment suspension

DETAILED DESCRIPTION:
Rationale A) primary endpoint

1. to verify the safety of protein sparing modified fast by enteral route ( EMF )in cycles of ten days/months repeated for six months,
2. To compare EMF with oral PSMF clinically ( appetite control, polmonary function tests and metabolic pattern) and on metabolic parameters (hypertension, glucose intolerance, dyslipidaemia) maintaining body composition (particularly fat free mass and muscular strength) in 15 patients with disease-causing obesity not responding to medical treatment and/or cognitive/behavioural therapy, who are candidates for invasive treatment such as the gastric balloon or surgery but do not intend to undergo them compared with 15 undergoing the same regimen without the naso-gastric tube. To verify the effects of treatment with regard to the enteral-hormonal structure during the acute phase (selected sub-group) and while undergoing treatment.

B) Secondary endpoints:

1. To verify the percentage of patients who maintain the weight reached 6 months after stopping treatment with the naso-gastric tube associated with a high-calorie normal-protein diet.
2. Verify clinical safety of EN in these patients.

ELIGIBILITY:
Inclusion Criteria:

* both genders, outpatients
* aged between 16 and 75
* with BMI 30 - 45 Kg/m2
* that are not in a restricted diet since at least 3 months
* with obesity related comorbidities (- type 2 diabetes
* mild or moderate OSAS
* orthopedic diseases (coxarthrosis, gonarthrosis)
* hypertension
* non alcoholic hepatic steatosis
* accepting to be enrolled in the study (signing informed consent)

Exclusion Criteria:

* Presence of gastrointestinal diseases
* Presence of cancer
* Patients treated with gastrolesive or anticoagulant drugs
* Hepatic failure, renal failure or multi-organ failure (cut off)
* Contraindications for enteral nutrition,Mechanical bowel complete, or partial chronic obstruction
* Severe mesenteric ischemia not caused by hypovolemia
* Digiunal or ileal fistula with high output (400 mL/die)
* Severe modifications of the intestinal function caused by enteropathies or insufficient absorbent surface, to the point that a normal nutritional state cannot be maintained
* Type 1 diabetes
* Type 2 diabetes treated with oral or injected drugs that may cause hypoglycemia
* ANBN: anorexia or bulimia nervosa, evaluation of other symptoms by specific tests
* Patients with major psychiatric disorders or not cooperative, or with alcohol or drug addiction disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with BMI 30 - 45 Kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-03-10 (Actual); Primary Completion 2012-12-20 (Actual); Study Completion 2012-12-20 (Actual)

PRIMARY OUTCOMES:
PSMF by tube feeding side effects | at the day 10th /month for 6 months
  Evaluation of side effects due to enteral nutrition by tube with a PSMF in obese subjects

CONTACTS AND LOCATIONS:
Overall Officials: Samir G Sukkar, MD, Study Director — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (1):
- IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy, Genova, Italy